CLINICAL TRIAL: NCT02740569
Title: Obstructive Sleep Apnea in Scleroderma and Pulmonary Involvement
Acronym: OSASPI
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2016.208
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Scleroderma, Systemic; Sleep Apnea, Obstructive; Pulmonary Disease
Keywords: scleroderma; sleep apnea; pulmonary disease
MeSH Terms: conditions — Scleroderma, Systemic; Sleep Apnea, Obstructive; Lung Diseases; Scleroderma, Diffuse; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for metabolic and cardiovascular markers
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — Observational study. Intervention according to the clinical routines (not included in this part)

SUMMARY:
Scleroderma is an autoimmune disease with skin manifestations and may have pulmonary involvement. Obstructive sleep apnea (OSA) may also be seen in scleroderma. Less is known regarding the prevalence of OSA in scleroderma and its association with pulmonary involvement.

DETAILED DESCRIPTION:
Scleroderma is an autoimmune disease with skin manifestations and may have pulmonary involvement. OSA may also be seen in scleroderma. Less is known regarding the prevalence of obstructive sleep apnea in scleroderma and its association with pulmonary involvement.

The investigators would like to address the prevalence of OSA in patients with Scleroderma, using overnight cardiorespiratory polygraphy. Other comorbidities and pulmonary findings on computer tomography (CT) as well as lung function tests will be evaluated.

The investigators plan to include 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Known scleroderma diagnosis
* Must be able to give informed consent

Exclusion Criteria:

* Serious neurological and/or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with known Scleroderma
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of OSA defined by apnea-hypopnea index (AHI) of at least 15/h on the overnight sleep study | 6 months
  All participants will be evaluated within 6 months

SECONDARY OUTCOMES:
Occurrence of pulmonary involvement based on computer tomography findings | 6 months
  All patients will be evaluated within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuksel Peker, MD, Prof, Principal Investigator — Marmara University Medical School
Locations (1):
- Marmara University, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yakut T, Balcan B, Karakurt S, Direskeneli H, Yalcinkaya Y, Peker Y. Impact of concomitant obstructive sleep apnea on pulmonary involvement and main pulmonary artery diameter in adults with scleroderma. Sleep Breath. 2021 Mar;25(1):135-143. doi: 10.1007/s11325-020-02059-4. Epub 2020 Apr 13. PMID 32285251